CLINICAL TRIAL: NCT07356895
Title: The Effect of the Social Stories Technique on Anesthesia Compliance in Children With Autism Spectrum Disorder
Brief Title: Effect of Social Stories on Anesthesia Compliance in Children With Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Sule Ozdemir, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AEŞH-EK-2025-311
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder; Social Stories
Keywords: Autism Spectrum Disorder; Social Stories; Preoperative Anxiety
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Stories Group (Active Comparator): Participants in this arm will receive the Social Stories Technique as a behavioral preoperative preparation intervention. Following informed consent, families will be provided with age- and developmentally appropriate Social Stories materials describing the anesthesia and surgical process using simple language and visual supports. Parents will be instructed to review the Social Stories with their child once daily.
  Interventions: Behavioral: Social Stories Group
- Routine Preoperative Preparation Group (Active Comparator): Participants in this arm will receive standard preoperative information as routinely provided in clinical practice. This includes verbal explanation of the anesthesia and surgical process given to the child's caregivers during the preoperative anesthesia consultation. No Social Stories materials or additional behavioral preparation tools will be provided.
  Interventions: Behavioral: Routine Preoperative Preparation Group

INTERVENTIONS:
Behavioral: Social Stories Group — The Social Stories Technique is a non-pharmacological behavioral intervention designed to prepare children with Autism Spectrum Disorder for anesthesia. Social Stories materials will be provided to families and will be read to the child by caregivers once daily for 7-14 days prior to surgery. The effect of the intervention on reducing preoperative anxiety and on cooperation during anesthesia induction-specifically compliance with intravenous cannulation and/or face mask application-will be evaluated.
  Arms: Social Stories Group
Behavioral: Routine Preoperative Preparation Group — Routine preoperative care consists of standard verbal information provided to caregivers regarding the anesthesia and surgical process during the preoperative anesthesia consultation. No Social Stories materials or additional behavioral preparation interventions will be used. Preoperative anxiety and cooperation during anesthesia induction, including compliance with intravenous cannulation and/or face mask application, will be evaluated.
  Arms: Routine Preoperative Preparation Group

SUMMARY:
Children with Autism Spectrum Disorder (ASD) frequently experience heightened anxiety and reduced cooperation during the perioperative period, which can complicate anesthesia induction and negatively affect procedural safety and efficiency. Non-pharmacological behavioral preparation methods that enhance predictability and understanding of medical procedures may improve anesthesia-related cooperation in this vulnerable population. The Social Stories Technique is a structured, visual-based behavioral intervention designed to support children with ASD by explaining upcoming experiences in a clear and developmentally appropriate manner.

This prospective controlled study aims to evaluate the effect of the Social Stories Technique on anesthesia compliance and preoperative anxiety in children with Autism Spectrum Disorder undergoing elective surgery. Children in the intervention group will receive Social Stories materials to be reviewed with their families prior to surgery, while the control group will receive standard preoperative information only. Primary and secondary outcomes will include anesthesia induction compliance, preoperative anxiety levels. The findings of this study are expected to contribute evidence regarding the effectiveness of a low-risk, non-pharmacological behavioral intervention to improve perioperative care in children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with Autism Spectrum Disorder
* Patients scheduled for elective surgical procedures
* Children aged 3 to 18 years
* American Society of Anesthesiologists (ASA) physical status class I-II
* Written informed consent obtained from a parent or legal guardian
* Caregivers willing and able to read the Social Stories materials at home as instructed
* Caregivers able to understand the Social Stories materials prepared in the Turkish language

Exclusion Criteria:

* Children with ASA physical status class III or higher systemic disease
* Patients requiring emergency surgery
* Children with severe intellectual disability or significant visual or hearing impairment
* History of severe behavioral problems during previous general anesthesia
* Families unable or unwilling to comply with the Social Stories intervention during the study period
* Inability to obtain written informed consent from a parent or legal guardian
* Children receiving pharmacological treatment for a comorbid psychiatric disorder

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2026-08-03 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Anesthesia Induction Compliance | During anesthesia induction on the day of surgery.
  Behavioral cooperation during anesthesia induction in children with Autism Spectrum Disorder will be assessed by compliance with face mask application and/or intravenous cannulation using the Induction Compliance Checklist (ICC).

SECONDARY OUTCOMES:
Preoperative Anxiety Level | Preoperative period on the day of surgery.
  Preoperative anxiety will be assessed using the Modified Yale Preoperative Anxiety Scale (mYPAS).
  The mYPAS is a validated observational scale evaluating preoperative anxiety across five behavioral domains (activity, vocalization, emotional expressivity, interaction with parents, and movement).
  Total scores range from 0 to 100, with higher scores indicating greater levels of preoperative anxiety.
  Clinically significant anxiety is generally considered at mYPAS scores ≥30-40.
Postoperative Agitation / Emergence Delirium | Immediate postoperative period in the post-anesthesia care unit.
  Postoperative agitation and emergence delirium will be assessed using the Pediatric Anesthesia Emergence Delirium (PAED) Scale.
  The PAED scale consists of five items scored from 0 to 4, yielding a total score ranging from 0 to 20.
  Higher PAED scores indicate more severe emergence delirium, and a total score of ≥10 is generally accepted as clinically significant emergence delirium.
Parental Satisfaction | On the day of surgery.
  Parental satisfaction with the perioperative process will be assessed using a 5-point Likert-type satisfaction scale, ranging from 1 (not satisfied at all) to 5 (very satisfied).
  Higher scores indicate greater parental satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)